CLINICAL TRIAL: NCT05282043
Title: Impacts of COVID-19 on Functional Capacity, Respiration, Pain, Depression, Sleep and Quality of Life on Young Adults
Brief Title: Pulmonary and Extrapulmonary Impacts of COVID-19 on Young Adults
Acronym: PEPICov
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, NAZLI GÜNGÖR, Lecturer, Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Istanbul Arel University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: PEPICov
Record Dates: First submitted 2022-03-13; First posted 2022-03-16 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Post COVID-19
Keywords: COVID-19; respiration; physical capacity; sleep; muscle strength; 6-minute walking test
MeSH Terms: conditions — COVID-19; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- post COVID-19 group (Experimental): In this group cases, who were infected with COVID-19 and had at least 12 weeks after diagnosis, will be allocated. Those should have no symptoms of COVID-19 such as fever, cough, ageusia, anosmia, diarrhea, arthralgia, myalgia, sore throat, headache, chest pain.
  Interventions: Other: Evaluation of Pulmonary and Extrapulmonary Impacts of COVID-19 on Young Adults
- healthy control group (Active Comparator): In this group cases, who were not infected with COVID-19 will be allocated.
  Interventions: Other: Evaluation of Pulmonary and Extrapulmonary Impacts of COVID-19 on Young Adults

INTERVENTIONS:
Other: Evaluation of Pulmonary and Extrapulmonary Impacts of COVID-19 on Young Adults — Participants' upper extremity and lower extremity muscle strength, 6-minute walking distance, O2 saturation, posture evaluation, spirometric evaluation, pain threshold, pain intensity, dyspnea, and leg fatigue measurements will be recorded. In addition to these measurements, general fatigue, quality of life, depression, physical activity level, sleep quality parameters will be evaluated and the data obtained will be analyzed with appropriate statistical methods.

SUMMARY:
When the literature search is conducted, it is seen that there are many studies examining the effects of COVID-19 disease on individuals in various disease groups (MS, stroke, Parkinson, COPD, asthma, etc.) and age groups (adult, geriatric, etc.). However, it has been determined that there is no study examining the impacts of this disease on functional capacity, physical activity, pulmonary function, emotional state, sleep, and quality of life in healthy young adults. This study will reveal whether COVID-19 disease causes an effect on the mentioned parameters in young adults. The aim of recent study is to investigate functional capacity, respiration, pain, depression, sleep and quality of life in young adults post COVID-19. For this purpose, participants' upper extremity and lower extremity muscle strength, 6-minute walking distance, O2 saturation, posture evaluation, spirometric evaluation, pain threshold, pain intensity, dyspnea, and leg fatigue measurements will be recorded. In addition to these measurements, general fatigue, quality of life, depression, physical activity level, sleep quality parameters will be evaluated and the data obtained will be analyzed with appropriate statistical methods.

The goals of recent work,

* To determine whether COVID-19 disease causes a decrease in functional capacity and changes in respiratory parameters in young adults, as well as to determine whether there are effects such as pain, depression, decreased sleep and quality of life,
* To determine whether there are significant changes in the values of the relevant outcome measurements in all the mentioned parameters,
* As a result of these, to determine the effects of COVID-19 disease on these parameters in young adults with objective, measurable data and to guide researchers and clinicians who do/will conduct studies on the subject.

ELIGIBILITY:
Inclusion Criteria:

* volunteers who are aged between 18-45 years
* cases, who were infected with COVID-19 and had at least 12 weeks after diagnosis
* cases, who have no symptoms of COVID-19 such as fever, cough, ageusia, anosmia, diarrhea, arthralgia, myalgia, sore throat, headache, chest pain

Exclusion Criteria:

* those have any cardiac or pulmonary disease history
* those have diagnoses of any psychological disease (major depression, anxiety disorder, etc.)
* those have any neurological or orthopaedic disease which hinders participation in physical activity

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2025-04-05 (Actual)

PRIMARY OUTCOMES:
6-minute walk test | up to 6 months
  unit: meters

SECONDARY OUTCOMES:
magnitude of muscle strength of upper and lower extremity | up to 6 months
  unit: Newtons
value of O2 saturation | up to 6 months
  unit: percent
Corbin's postural assessment | up to 6 months
  This scale has a total score range between 0-18. Every subscore range refers to specific situations about posture. These are mentioned below:
  0-4: Excellent 5-7: Very good 8-10: Good 11-13: Fair 14 or more: Poor
spirometer testing | up to 6 months
  FEV1, FVC, FEV1/FVC values
pressure pain threshold | up to 6 months
  unit: Newtons/cm2
pain intensity | up to 6 months
  unit: millimeters (according to Visual Analog Scale)
dyspnea severity | up to 6 months
  (according to Modified Borg Scale) This scale has a total score range between 0-10. Every subscore refers to specific situations about dyspnea. These are mentioned below: 0: No Exertion 0.5: Very very Slight
  1. Very Slight
  2. Slight
  3. Moderate
  4. Somewhat Severe
  5. Severe 6
  7: Very Severe 8 9: Very very Severe 10: Maximal
leg fatigue | up to 6 months
  (according to Modified Borg Scale) This scale has a total score range between 0-10. Every subscore refers to specific situations about leg fatigue. These are mentioned below: 0: No Exertion 0.5: Very very Slight
  1. Very Slight
  2. Slight
  3. Moderate
  4. Somewhat Severe
  5. Severe 6
  7: Very Severe 8 9: Very very Severe 10: Maximal
general fatigue | up to 6 months
  (according to Fatigue Severity Scale) This scale has a 9-item which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients. Its minimum value is 9 and the maximum is 63. The higher the score indicates more severe fatigue and more impact on the person's activities.
quality of life questionnaire | up to 6 months
  (according to Short Form-36) This form contains 36 questions. There are 8 different parameters of the questionnaire. These are mentioned below:
  * Physical functioning
  * Role limitations due to physical health
  * Role limitations due to emotional problems
  * Energy/fatigue
  * Emotional well-being
  * Social functioning
  * Pain
  * General health Every parameter has an average score that ranges between 0-100. Higher score indicates better situations that are specific to every parameter.
depression severity | up to 6 months
  (according to Beck Depression Inventory) This inventory has a score range between 0-63. Certain score ranges refer to specific conditions. These are mentioned below: 1-10: normal 11-16: Mild mood disturbance 17-20: Borderline clinical depression 21-30: Moderate depression 31-40: Severe depression over 40: Extreme depression
physical activity level (according to International Physical Activity Questionnaire/short form) | up to 6 months
  In this form, there are 4 different activities which have a certain MET level. The formule which is used for obtain a total score is presented below:
  -MET level x minutes of activity x events per week
  According to total score, a classification is established:
  Inactive
  * No activity OR
  * Some activity but not enough to meet Categories 2 or 3. Minimally Active Any one of the following criterias
  * 3 or more days of vigorous activity of at least 20 minutes per day
  * 5 or more days of moderate intensity activity or walking of at least 30 minutes per day
  * 5 or more days of any combination of walking, moderate-intensity or vigorous activities achieving a minimum of at least 600 MET-min/week.
  HEPA active Any one of the following criterias
  * Vigorous-intensity activity on at least 3 days and accumulating at least 1500 MET-minutes/week
  * 7 or more days of any combination of walking, moderate-intensity or vigorous activities achieving a minimum of at least 3000 MET-minutes/week
quality of sleep | up to 6 months
  (according to Pittsburgh Sleep Quality Index) This index has 7 components and overall scoring alters between 0-21 points. 0 point indicates no difficulty while 21 points indicate severe difficulties.

OTHER OUTCOMES:
The post-COVID-19 functional status (PCFS) scale | up to 6 months
  The post-COVID-19 functional status (PCFS) scale focuses on relevant aspects of daily life during follow-up after the infection. The scale is intended to help users becoming aware of current functional limitations in COVID-19 patients, whether or not as a result of the specific infection, and to objectively determine this degree of disability. As such, the scale is not meant to replace other relevant instruments for measuring quality of life, tiredness or dyspnoea, but is developed to use as an additional tool for evaluating the ultimate consequences of COVID-19 on functional status. The scale is ordinal, has 6 steps ranging from 0 (no symptoms) to 5 (death, D), and covers the entire range of functional outcomes by focusing on limitations in usual duties/activities either at home or at work/study, as well as changes in lifestyle.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Arel University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tuzun S, Keles A, Okutan D, Yildiran T, Palamar D. Assessment of musculoskeletal pain, fatigue and grip strength in hospitalized patients with COVID-19. Eur J Phys Rehabil Med. 2021 Aug;57(4):653-662. doi: 10.23736/S1973-9087.20.06563-6. Epub 2021 Jan 4. PMID 33393277
- [Result] Lee CC, Wu HJ, Chiou WB. Reminders of COVID-19 social distancing can intensify physical pain. Br J Soc Psychol. 2022 Apr;61(2):587-598. doi: 10.1111/bjso.12498. Epub 2021 Sep 12. PMID 34510481
- [Result] Tanriverdi A, Savci S, Kahraman BO, Ozpelit E. Extrapulmonary features of post-COVID-19 patients: muscle function, physical activity, mood, and sleep quality. Ir J Med Sci. 2022 Jun;191(3):969-975. doi: 10.1007/s11845-021-02667-3. Epub 2021 Jun 2. PMID 34080125